CLINICAL TRIAL: NCT06783907
Title: Technological-based Personalized Care Intervention for Supporting Older People With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Queenie Law Pui Sze, Associate Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HE-RD/2023/1.11
Record Dates: First submitted 2024-12-12; First posted 2025-01-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive technology for continuous glucose monitoring; Diabetes Mellitus Self-management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non invasive blood glucose monitoring group (Experimental): Non invasive blood glucose monitoring : Participants will use a non-invasive sensor on the arm for blood glucose monitoring during the first and second weeks, as well as the seventh and eighth weeks. Between the third and sixth weeks, participants will be asked to monitor their blood glucose levels at home using traditional methods.
  Interventions: Behavioral: Non-invasive blood glucose monitoring
- Traditional blood glucose monitoring (Active Comparator): Traditional blood glucose monitoring : Participants will engage in traditional self-monitoring of blood glucose at home over the course of 8 weeks. They are recommended to check their blood glucose levels one to two times per week and record all results. This will allow for the collection of data using traditional monitoring methods.
  Interventions: Behavioral: Traditional blood glucose monitoring

INTERVENTIONS:
Behavioral: Non-invasive blood glucose monitoring — Non-invasive wearable glucose monitoring device for capturing participants' blood glucose.
  The intervention will include:
  1. Training for self-management of diabetes and phone consultation.
  2. Follow-up through phone calls or WhatsApp for hypoglycaemic or hyperglycaemic events.
  3. Personalized care guided by sensor data.
  The Investigator will monitor the health data from the device regularly. A mobile app will track and record compliance with blood glucose monitoring.
  Arms: Non invasive blood glucose monitoring group
Behavioral: Traditional blood glucose monitoring — Traditional blood glucose monitoring
  Participants will engage in traditional self-monitoring of blood glucose at home over the course of 8 weeks. They are recommended to check their blood glucose levels one to two times per week and record all results. This will allow for the collection of data using traditional monitoring methods.
  Arms: Traditional blood glucose monitoring

SUMMARY:
The objectives of this project are (1) to develop a new model of DM management using non-invasive healthcare technology for continuous glucose monitoring; (2) to use health apps to give timely personalized care intervention for enhancing compliance rate of DM self-management; & (3) to compare the DM management using non-invasive healthcare technology to traditional invasive blood glucose monitoring method.

The proposed study will adopt a RCT with two treatment arms to clarify the effects of non-invasive blood glucose device on blood glucose monitoring. The two arms will be the non-invasive blood glucose monitoring (arm 1) and traditional self-monitoring (arm 2) as a control. A block randomisation and a single-blind design will be used. The inclusion criteria are (1) aged ≥ 60 years old; (2) patients diagnosed with Type II DM; (3) patients experienced hypo (histix < 4.0 mmol/L) or hyperglycemia (histix ≥16.0 mmol/L); & (iv) the Abbreviated Mental Test (AMT) ≥ 6.

Participants fitting the inclusion criteria will be selected by convenience sampling. They will join a two-arm RCT and will be allocated into the intervention or control group in a 1:1 ratio.

The primary outcomes will be the point of care test (POCT) of HbA1C level and the secondary outcomes will be the fasting blood glucose, total cholesterol, blood pressure, basic anthropometric measurement, breath and blood ketone and Diabetes Self-Care activities questionnaire. The outcome measurements will be recorded before the intervention (T0) and immediately after the 8-week intervention (T1).

The required sample size would be 30 participants per group (with a ratio of 1:1) for testing the feasibility of the study.

DETAILED DESCRIPTION:
Research aim

1. This study will aim to develop a new model of DM management using non- invasive healthcare technology for continuous glucose monitoring.

2 To use health apps to give timely personalized care intervention for enhancing compliance rate of DM self-management. 3. To compare the DM management using non-invasive healthcare technology to traditional invasive blood glucose monitoring method. 4. To improve self-management skills, decrease hospital admissions, and save medical.

Our DM project integrates personalized care intervention with a non-invasive continuous glucose monitoring (CGM) device for diabetes patients. The use of mHealth (Mobile health) ensures timely care without time or location constraints, while Just-in-Time Adaptive Intervention (JITAI) provides instant, personalized support. The painless, non-invasive CGM device offers an alternative to traditional finger-prick methods, improving compliance with self-management. This approach is particularly beneficial for patients who struggle with conventional monitoring and aims to enhance both patient outcomes and healthcare efficiency, especially for older people at high risk of hypo- or hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 60 years old;
2. patients diagnosed with Type II DM without insulin injections;
3. patients experienced hypo (histix < 4.0 mmol/L) or hyperglycemia (histix

   * 16.0 mmol/L); &

2. The Abbreviated Mental Test (AMT) ≥ 6.

Exclusion Criteria:

1. patient on dialysis;
2. taking ascorbic acid > 500mg daily or (Not recommended by manufacturer as result may be affected);
3. taking salicylic acid ≥ 650mg single dose or (Not recommended by manufacturer as result may be affected); or
4. scheduled radiological therapy during CGM application (Not recommended by manufacturer as result may be affected).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
The point of care test (POCT) of HbA1C level | 8 weeks
  Change in HbA1C level The HbA1C will be measured by A1CNow system.

SECONDARY OUTCOMES:
Change in lipid and glucose panel | 8 weeks
  Change in lipid and glucose panel measured by CardioChek
Change in basic anthropometric measurement | 8 weeks
  Change in basic anthropometric measurement:
  1. Height will be measured in meters using a tape measure.
  2. Weight will be measured in kilograms using a scale.
  3. Weight and height will be combined to report Body Mass Index (BMI) in kg/m^2
Change in blood pressure | 8 weeks
  Change in blood pressure:
  Measured using Omron M7 blood pressure monitors to assess brachial blood pressure
Change in breath and blood ketone | 8 weeks
  Change in breath and blood ketone:
  Used to detect ketones in the breath and blood, indicating hyperglycemia or diabetic ketoacidosis in individuals with diabetes
Change in Summary of Diabetes Self-Care Activities (SDSCA) Chinese Version | 8 weeks
  Change in Summary of Diabetes Self-Care Activities (SDSCA) Chinese Version:
  Used to assess participants' diabetes self-care activities.

CONTACTS AND LOCATIONS:
Locations (1):
- LEI FOOK Neighbourhood Elderly Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] 2. World Health Organization. (2016). Global Report on Diabetes. In World Health Organization (Vol. 978). https://doi.org/ISBN 978 92 4 156525 7
- [Background] 3. Centre for Health Protection. (2017). Report of Population Health Survey 2014/2015.
- [Background] Wang L, Miller LC. Just-in-the-Moment Adaptive Interventions (JITAI): A Meta-Analytical Review. Health Commun. 2020 Nov;35(12):1531-1544. doi: 10.1080/10410236.2019.1652388. Epub 2019 Sep 5. PMID 31488002
- [Background] Goldstein SP, Zhang F, Klasnja P, Hoover A, Wing RR, Thomas JG. Optimizing a Just-in-Time Adaptive Intervention to Improve Dietary Adherence in Behavioral Obesity Treatment: Protocol for a Microrandomized Trial. JMIR Res Protoc. 2021 Dec 6;10(12):e33568. doi: 10.2196/33568. PMID 34874892
- [Background] Hardeman W, Houghton J, Lane K, Jones A, Naughton F. A systematic review of just-in-time adaptive interventions (JITAIs) to promote physical activity. Int J Behav Nutr Phys Act. 2019 Apr 3;16(1):31. doi: 10.1186/s12966-019-0792-7. PMID 30943983
- [Background] Teepe GW, Da Fonseca A, Kleim B, Jacobson NC, Salamanca Sanabria A, Tudor Car L, Fleisch E, Kowatsch T. Just-in-Time Adaptive Mechanisms of Popular Mobile Apps for Individuals With Depression: Systematic App Search and Literature Review. J Med Internet Res. 2021 Sep 28;23(9):e29412. doi: 10.2196/29412. PMID 34309569
- [Background] Perski O, Hebert ET, Naughton F, Hekler EB, Brown J, Businelle MS. Technology-mediated just-in-time adaptive interventions (JITAIs) to reduce harmful substance use: a systematic review. Addiction. 2022 May;117(5):1220-1241. doi: 10.1111/add.15687. Epub 2021 Oct 11. PMID 34514668
- [Background] 9. Pimenta, N., Félix, I. B., Monteiro, D.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT06783907/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT06783907/ICF_001.pdf